CLINICAL TRIAL: NCT00330681
Title: A Confirmatory Study of MCI-186 for Treatment of Amyotrophic Lateral Sclerosis in Double-blind, Parallel-group, Placebo-controlled Manner.
Brief Title: Efficacy and Safety Study of MCI-186 for Treatment of Amyotrophic Lateral Sclerosis (ALS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MCI186-16
Record Dates: First submitted 2006-05-26; First posted 2006-05-29 (Estimated); Results first posted 2017-05-17 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
Keywords: Amyotrophic lateral sclerosis; free radical scavenger
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Edaravone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): MCI-186
  Interventions: Drug: MCI-186
- 2 (Placebo Comparator): Placebo of MCI-186
  Interventions: Drug: Placebo of MCI-186

INTERVENTIONS:
Drug: MCI-186 — Two ampoules (60 mg) of MCI-186 injection are intravenously administered once a day, for successive 14 days, followed by 14 days observation period (first cycle). Then treatment (10 days' administration during 14 days) - observation (14 days) cycle is repeated five times (2nd-6th cycles).
  Other Names: Edaravone; Radicut
  Arms: 1
Drug: Placebo of MCI-186 — Two ampoules of placebo injection are intravenously administered once a day, for successive 14 days, followed by 14 days observation period (first cycle). Then treatment (10 days' administration during 14 days) - observation (14 days) cycle is repeated five times (2nd-6th cycles).
  Arms: 2

SUMMARY:
The primary objective of this study is to confirm the efficacy of 60 mg of MCI-186 via intravenous drip once a day in patients with ALS based on the changes in the revised ALS functional rating scale (ALSFRS-R) scores after 24 weeks administration in double-blind, placebo-controlled manner. And in addition, this study will be performed to examine the safety of MCI-186 to ALS patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are defined as "definite ALS," "probable ALS" or "probable-laboratory-supported ALS," met diagnostic criteria revised EL Escorial for Airlie House.
* Patients who can eat a meal, excrete, or move with oneself alone, and do not need assistance in everyday life.
* Patients of less than 3 years after the onset of ALS.
* Patients whose progress of the condition during 12 weeks before administration meet other requirements.

Exclusion Criteria:

* Patients judged to be inadequate to participate in this study by their physician, because those patients' general condition deteriorated to the point that they need to be hospitalized for severe hepatic disease, severe heart disease, severe renal disease and so on, or they need to be administered antibiotics to infection.
* Patients who complain the difficulty in breathing caused by deteriorating the respiratory function.
* Patients with such complications as Parkinson's disease, schizophrenia, dementia, renal failure, or other severe complication, and patients who have the anamnesis of hypersensitivity to edaravone.
* Pregnant, lactating, and probably pregnant patients, and patients who want to become pregnant, and patients who can not agree to contraception.
* Patients who have participated in other trials within 12 weeks before consent, or who are participating in other clinical trials at present.
* In addition to the above exclusion criteria, patients judged to be inadequate to participate in this study by their physician.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2006-05; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Koji Abe, professor, Study Chair — Graduate School of Medicine and Dentistry, Okayama University

REFERENCES:
- [Result] Abe K, Itoyama Y, Sobue G, Tsuji S, Aoki M, Doyu M, Hamada C, Kondo K, Yoneoka T, Akimoto M, Yoshino H; Edaravone ALS Study Group. Confirmatory double-blind, parallel-group, placebo-controlled study of efficacy and safety of edaravone (MCI-186) in amyotrophic lateral sclerosis patients. Amyotroph Lateral Scler Frontotemporal Degener. 2014 Dec;15(7-8):610-7. doi: 10.3109/21678421.2014.959024. Epub 2014 Oct 6. PMID 25286015

RESULTS

PARTICIPANT FLOW:
Groups:
- MCI-186: Edaravone 60 mg, intravenously infused over 60 min once daily.
- Placebo of MCI-186: Edaravone matched placebo, intravenously infused over 60 min once daily.
Period: Overall Study
Arm/Group | MCI-186 | Placebo of MCI-186
Started | 102 | 104
Completed | 93 | 90
Not Completed | 9 | 14
Not completed — Adverse Event | 3 | 6
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 5 | 5
Not completed — Tracheotomy due to worsening of ALS | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MCI-186 | Placebo of MCI-186 | Total
Number analyzed (Participants) | 102 | 104 | 206
Age, Customized [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 19 and 64 years | 74 | 71 | 145
  >=65 years | 28 | 33 | 61
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 35 | 73
  Male | 64 | 69 | 133

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Revised ALS Functional Rating Scale (ALSFRS-R) Score in Full Analysis Set (FAS) Population at 24 Weeks
Description: ALSFRS-R Score: 0=worst; 48=best
Time Frame: baseline and 24 weeks
Population: "1 patient with diseases other than ALS" and "1 patient who did not reach the end of cycle 3" were excluded from the FAS in the MCI-186 group.
  "5 patients who did not reach the end of cycle 3" were excluded from the FAS in the Placebo of MCI-186 group.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | MCI-186 | Placebo of MCI-186
Number analyzed (Participants) | 100 | 99
units on a scale | -5.7 (0.85) | -6.35 (0.84)

2. Secondary Outcome: Death or a Specified State of Disease Progression
Description: Any of "death, disability of independent ambulation, loss of upper arm function, tracheotomy, use of respirator, and use of tube feeding" was defined as an event.
Time Frame: 24 weeks
Population: "1 patient with diseases other than ALS" was excluded from the FAS in the MCI-186 group.
Measure: Number; unit: participants
Arm/Group | MCI-186 | Placebo of MCI-186
Number analyzed (Participants) | 101 | 104
participants
  death | 2 | 2
  disability of independent ambulation | 28 | 23
  loss of upper arm function | 2 | 4
  tracheotomy | 0 | 2
  use of respirator | 1 | 3
  use of tube feeding | 5 | 3

3. Secondary Outcome: Change From Baseline in % Forced Vital Capacity (%FVC) in Full Analysis Set (FAS) Population at 24 Weeks
Time Frame: baseline and 24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of FVC
Arm/Group | MCI-186 | Placebo of MCI-186
Number analyzed (Participants) | 100 | 99
percentage of FVC | -14.57 (2.41) | -17.49 (2.39)

4. Secondary Outcome: Change From Baseline in Modified Norris Scale Score in Full Analysis Set (FAS) Population at 24 Weeks
Description: The Modified Norris Scale is a measure of movement disorder for patients with ALS. Worst=0, Best=102
Time Frame: baseline and 24 weeks
Population: "1 patient with diseases other than ALS", "1 patient who did not reach the end of cycle 3" and "5 patients with missing data" were excluded from the FAS in the MCI-186 group.
  "5 patients who did not reach the end of cycle 3" and "2 patients with missing data" were excluded from the FAS in the Placebo of MCI-186 group.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | MCI-186 | Placebo of MCI-186
Number analyzed (Participants) | 95 | 97
units on a scale | -14.12 (2.05) | -16.15 (2)

5. Secondary Outcome: Change From Baseline in ALS Assessment Questionnaire (40 Items) (ALSAQ40) in Full Analysis Set (FAS) Population at 24 Weeks
Description: The ALSAQ40 score is a measure of QoL for patients with ALS. The ALSAQ40 evaluates domains that include physical mobility, ADL and independence, eating and drinking, communication, and emotional reactions. Worst=200, Best=40
Time Frame: baseline and 24 weeks
Population: "1 patient with diseases other than ALS", "1 patient who did not reach the end of cycle 3" and "5 patients with missing data" were excluded from the FAS in the MCI-186 group.
  "5 patients who did not reach the end of cycle 3" and "4 patients with missing data" were excluded from the FAS in the Placebo of MCI-186 group.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | MCI-186 | Placebo of MCI-186
Number analyzed (Participants) | 95 | 95
units on a scale | 19.6 (3.82) | 19.13 (3.79)

6. Secondary Outcome: Percentage of Participants With Adverse Events
Time Frame: 24 weeks
Measure: Number; unit: percentage of participants
Arm/Group | MCI-186 | Placebo of MCI-186
Number analyzed (Participants) | 102 | 104
percentage of participants | 89.2 | 88.5

7. Secondary Outcome: Percentage of Participants With Adverse Drug Reactions
Time Frame: 24 weeks
Measure: Number; unit: percentage of participants
Arm/Group | MCI-186 | Placebo of MCI-186
Number analyzed (Participants) | 102 | 104
percentage of participants | 13.7 | 19.2

8. Secondary Outcome: Percentage of Participants With Laboratory Tests for Which the Incidence of Abnormal Changes Was 5% or Higher in Either Group
Time Frame: 24 weeks
Population: "1 patient with missing data" was excluded from the FAS in the Placebo of MCI-186 group.
Measure: Number; unit: percentage of participants
Arm/Group | MCI-186 | Placebo of MCI-186
Number analyzed (Participants) | 102 | 103
percentage of participants
  White blood cell count | 2 | 5.8
  urinary glucose | 6.9 | 2.9

9. Secondary Outcome: Percentage of Participants With Abnormal Changes in Sensory Examinations
Time Frame: 24 weeks
Measure: Number; unit: percentage of participants
Arm/Group | MCI-186 | Placebo of MCI-186
Number analyzed (Participants) | 102 | 104
percentage of participants
  Numbness | 1 | 1
  Staggering | 2 | 3.8
  Vibratory sensation | 0 | 1

ADVERSE EVENTS:
Arm/Group | MCI-186 | Placebo of MCI-186
Serious Adverse Events (participants affected / at risk) | 18/102 | 24/104
Other Adverse Events (participants affected / at risk) | 88/102 | 91/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MCI-186 (N=102) | Placebo of MCI-186 (N=104)
Vertigo positional (Ear and labyrinth disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 8 | 11
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Abasia (General disorders) | 1 | 0
Gait disturbance (General disorders) | 3 | 2
Oedema peripheral (General disorders) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 1
Mastication disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 3 | 3
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dyslalia (Nervous system disorders) | 1 | 2
Anxiety (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MCI-186 (N=102) | Placebo of MCI-186 (N=104)
Anaemia (Blood and lymphatic system disorders) | 0 | 3
Palpitations (Cardiac disorders) | 1 | 0
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0
Cerumen impaction (Ear and labyrinth disorders) | 1 | 0
Eustachian tube patulous (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 2
Vertigo positional (Ear and labyrinth disorders) | 1 | 1
Astigmatism (Eye disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 2
Conjunctivitis (Eye disorders) | 1 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 1
Dry eye (Eye disorders) | 1 | 0
Eye discharge (Eye disorders) | 0 | 1
Eye pain (Eye disorders) | 1 | 1
Eye pruritus (Eye disorders) | 0 | 1
Myodesopsia (Eye disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Anal prolapse (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 13 | 17
Dental caries (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 5
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 2 | 2
Gingival swelling (Gastrointestinal disorders) | 0 | 1
Gingivitis (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1
Periodontitis (Gastrointestinal disorders) | 1 | 0
Sensitivity of teeth (Gastrointestinal disorders) | 1 | 0
Stomach discomfort (Gastrointestinal disorders) | 0 | 2
Stomatitis (Gastrointestinal disorders) | 1 | 5
Tooth loss (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Abasia (General disorders) | 1 | 0
Catheter site erythema (General disorders) | 0 | 1
Catheter site inflammation (General disorders) | 0 | 2
Catheter site pain (General disorders) | 0 | 1
Chest pain (General disorders) | 2 | 0
Feeling abnormal (General disorders) | 1 | 1
Gait disturbance (General disorders) | 17 | 14
Infusion site reaction (General disorders) | 1 | 0
Injection site phlebitis (General disorders) | 0 | 1
Local swelling (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Oedema (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 3
Pyrexia (General disorders) | 1 | 1
Thirst (General disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 5
Hepatic steatosis (Hepatobiliary disorders) | 2 | 0
Liver disorder (Hepatobiliary disorders) | 2 | 0
Seasonal allergy (Immune system disorders) | 0 | 1
Bronchitis (Infections and infestations) | 2 | 3
Cystitis (Infections and infestations) | 2 | 2
Enterocolitis bacterial (Infections and infestations) | 0 | 1
Folliculitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 3
Herpes zoster (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 3 | 2
Nail infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 22 | 22
Onychomycosis (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0
Otitis externa (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 1 | 1
Pharyngitis (Infections and infestations) | 3 | 2
Pneumonia (Infections and infestations) | 0 | 1
Purulence (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 0 | 1
Tinea capitis (Infections and infestations) | 0 | 1
Tinea cruris (Infections and infestations) | 0 | 1
Tinea infection (Infections and infestations) | 1 | 0
Tinea pedis (Infections and infestations) | 2 | 1
Tonsillitis (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 1 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 2
Back injury (Injury, poisoning and procedural complications) | 1 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 12 | 5
Excoriation (Injury, poisoning and procedural complications) | 3 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 1
Joint sprain (Injury, poisoning and procedural complications) | 3 | 0
Open wound (Injury, poisoning and procedural complications) | 1 | 1
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 2
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 2
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 0 | 1
Blood urea increased (Investigations) | 1 | 0
Blood urine present (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Glucose urine present (Investigations) | 6 | 3
Liver function test abnormal (Investigations) | 1 | 0
Protein urine present (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 5
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6 | 8
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 2
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 2
Dizziness postural (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 8 | 3
Intercostal neuralgia (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Pallanaesthesia (Nervous system disorders) | 0 | 1
Post herpetic neuralgia (Nervous system disorders) | 1 | 0
Sensory disturbance (Nervous system disorders) | 0 | 1
Tension headache (Nervous system disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 9 | 10
Calculus urinary (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1
Nocturia (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Epididymitis (Reproductive system and breast disorders) | 0 | 1
Gynaecomastia (Reproductive system and breast disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Acrodermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 3 | 2
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 7 | 2
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 3
Erythema (Skin and subcutaneous tissue disorders) | 3 | 2
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 1 | 0
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 2
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3
Purpura (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 4 | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1
Xeroderma (Skin and subcutaneous tissue disorders) | 1 | 0
Essential hypertension (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 2
Phlebitis (Vascular disorders) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other